CLINICAL TRIAL: NCT04543864
Title: Soft Tissue Changes Assessment in Screw-Retained Maxillary Implant Supported Complete Denture With Electric Welded Metal Framework Versus Casted One (RCT, Split Mouth Design)
Brief Title: Soft Tissue Assessment in Screw-Retained Maxillary Complete Denture With Electric Welded Framework Versus Casted
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hamsa Khalid Lafta, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13420
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electric welded metal framework (Experimental)
  Interventions: Device: Electric intraoral welding device
- conventional casted metal framework (Experimental)
  Interventions: Device: casting

INTERVENTIONS:
Device: Electric intraoral welding device — welding metal framework to the implants in completely edentulous maxilla by electric welding device intraorally
  Arms: electric welded metal framework
Device: casting — casting the metal framework
  Arms: conventional casted metal framework

SUMMARY:
comparing the changes in the soft tissue around the implants that will be joined by a metal framework either with electric welding or with the conventional casting method

DETAILED DESCRIPTION:
as joining multiple implants by a metal framework considered a solid solution for edentulous arches , but in the same time the conventional method to weld this metal framework to the implants by casting technique in lab usually involves a several disadvantages eg. cost and time consuming in addition to laboratory errors, Thus , this study aims to find another method to weld the metal framework intraorally by an electric welding device

ELIGIBILITY:
Inclusion Criteria:

* Ages range from 45 to 65 years old.
* Absence of any medical disorder that could complicate the Surgical phase or affect osseointegration.
* The patients must be completely edentulous.
* The patient must have enough bone height for implants minimum length of 10mm and a minimum diameter of 5 mm.
* Patients with good oral hygiene.
* Complete denture wearer.
* Adequate inter arch space for screw retained prosthesis.
* Absence of any intra-oral pathological condition.

Exclusion Criteria:

* Patients with recent extraction(less than three months).
* Patients with inflamed ridge or candida infection.
* Patients with flappy ridge.
* Parafunctional habits.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Soft Tissue Changes Assessment | 12 months
  Primary outcome is the probing depth which will be measured using the periodontal probe (unit mm) around the implant to check the changes that may occur in the peri-implant soft tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University , Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No